CLINICAL TRIAL: NCT04944264
Title: SMART Management of Type 1 Diabetes - Modifying Glucose Metabolism With an Online Mind-body Intervention: A Feasibility and Pilot Study
Brief Title: A Mind-Body Intervention for Diabetes Management: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, James E. Stahl, Associate Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02000298
Record Dates: First submitted 2021-06-09; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus; Stress, Psychological; Stress, Physiological
MeSH Terms: conditions — Diabetes Mellitus; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate start (Active Comparator): Behavioral: Stress Management and Resiliency Training (SMART) program
  Interventions: Behavioral: Stress Management and Resiliency Training (SMART) program
- Delayed start (Active Comparator): Wait time control
  Interventions: Behavioral: Stress Management and Resiliency Training (SMART) program

INTERVENTIONS:
Behavioral: Stress Management and Resiliency Training (SMART) program — The Stress Management and Resiliency Training (SMART) program (bensonhenryinstitute.org) is well validated comprehensive stress management program. It is designed to cultivate both the early recognition of stress in the mind and body, develop skills to mitigate stress and evoke the relaxation response and cultivate resiliency. It is an 8 session program, typically run in a live group setting. In this study's case it was delivered via a videoconferencing platform.

SUMMARY:
Managing type 1 diabetes is stressful. Stress physiology influences glucose metabolism. Continuous glucose monitors allow us to track glucose variability in the real-world environment. Managing stress and cultivating resiliency should improve diabetes management and reduce glucose variability. The study was designed as a randomized prospective cohort pre-post study with wait time control. Participants were adult type 1 diabetes patients who used a continuous glucose monitor and recruited from an academic endocrinology practice. The intervention was the Stress Management and Resiliency Training (SMART) program conducted over 8 sessions over web-based video conference software. The primary outcome measures were: Glucose variability, the Diabetes Self-Management questionnaire (DSMQ) and the Connor-Davidson Resiliency (CD-RISC) instrument.

DETAILED DESCRIPTION:
Hypothesis: It was hypothesized that the course on videoconferencing platform would deliver similar effects on quality of life as has been seen in the past from on-site courses, and that the intervention would reduce glucose variability and improve resiliency Design: This pilot was designed as a prospective cohort pre-post intervention study with subjects randomized to an immediate start or wait time control The study was approved by the Committee for the Protection of Human Subjects at Dartmouth Hitchcock Medical Center and Dartmouth College. All participants provided written informed consent.

Intervention: The Stress Management and Resiliency Training (SMART) program (bensonhenryinstitute.org) is well validated comprehensive stress management program. It is designed to cultivate both the early recognition of stress in the mind and body, develop skills to mitigate stress and evoke the relaxation response and cultivate resiliency. It is an 8 session program, typically run in a live group setting. In this study's case it was delivered via a videoconferencing platform. This was done both as a means of testing delivering this service in a rural setting where patient might be geographically distant or isolated and to accommodate the need for social distancing during the COVID-19 pandemic.

Recruitment: Recruitment occurred through the Dartmouth-Hitchcock Medical Center (DHMC) endocrinology clinic and the endocrinologists working there. Candidates were included if they had type 1 diabetes and used a continuous glucose monitor. Candidates were excluded if they were < 21 years old and could not give informed consent. To allow for controlled analysis, on presentation at each site, participants were randomly assigned to one of two cohorts: 1) immediate start (A) and 2) delayed start (B). The immediate arm began at the next available class. The delayed start group began 4 weeks later. During their wait, this group was offered usual care.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 1 diabetes (diagnosis ≥ 5 years) treated exclusively with insulin by multiple (>2 daily) injections or pump
* no prior use of a continuous glucose monitor; ages > 21
* ability to read and speak English at the high school level
* ability and willingness to come to the clinic once per week for a mind-body group intervention.

Exclusion Criteria:

* major psychiatric illness
* severe diabetes complications under active treatment (i.e., retinal laser or injection treatments, dialysis, foot ulcers)
* pregnancy
* an inability to attend weekly mind-body group sessions

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Glucose (mg/dl) | duration of study, approximately 6 months
  Glucose levels measured via a continuous glucose monitor (CGM) in order to determine Mean, Median and Standard Deviation over 10 days total for both sleep time (10 PM to 6 AM) and active time (6 AM to 10 PM); data is automatically collected every 15 minutes
Glucose standard deviation (SD) | duration of study, approximately 6 months
  Glucose levels measured via a continuous glucose monitor (CGM) in order to determine Mean, Median and Standard Deviation over 10 days total for both sleep time (10 PM to 6 AM) and active time (6 AM to 10 PM); data is automatically collected every 15 minutes
Glucose Management Indicator (GMI) | duration of study, approximately 6 months
  Glucose Management Indicator (GMI) approximates the laboratory A1C level expected based on average glucose measured using continuous glucose monitoring (CGM) values. Average glucose is derived from at least 12 days of CGM data
Short Form - 6 Dimensions (SF-6D) | duration of study, approximately 6 months
  Range 0 - 1. Higher is better an econometric preference-based index derived from 11 items of the SF-36, which are combined into six dimensions of health, with four to six levels each. It is used to estimate quality of life. The SF-6D describes 18,000 different health states.
Diabetes Self-Management Questionnaire (DSMQ) | duration of study, approximately 6 months
  Range 0 - 10. Higher is better The DSMQ is a 16-item questionnaire to assess self-care activities associated with glycemic control in patients with diabetes.
Connor-Davidson Resilience Scale (CD-RISC) | duration of study, approximately 6 months
  Range 0 - 25. Higher is better The CD-RISC assesses resilience and constitutes a 25 item questionnaire scored on a 5-point likert scale (rated 0-4). The total score ranges from 0-100, with higher scores indicating greater resilience.

SECONDARY OUTCOMES:
Implementation barriers | duration of study, approximately 6 months
  Qualitative feedback from participants regarding implementation barriers of the SMART-3RP program for patients with type 1 diabetes
Implementation Facilitators | duration of study, approximately 6 months
  Qualitative feedback from participants regarding Implementation Facilitators of the SMART-3RP program for patients with type 1 diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stahl JE, Ammana HR, Kwak L, Comi RJ. SMART-ly Managing Type 1 Diabetes - Modifying Glucose Metabolism With an Online Mind-Body Intervention: A Feasibility and Pilot Study. Front Clin Diabetes Healthc. 2022 Mar 3;3:802461. doi: 10.3389/fcdhc.2022.802461. eCollection 2022. PMID 36992749